CLINICAL TRIAL: NCT05648162
Title: Convergence of Acupuncture and Transcranial Direct Current Stimulation(tDCS) Rehabilitation Effect on Motor Function of Patients of Acute Stroke
Brief Title: Acupuncture-tDCS Convergence Rehabilitation Effect on Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-2022-002
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical acupuncture+ tDCS + NDT-Bobath Rehabilitation (Experimental): Electrical acupuncture, tDCS, and NDT-BOBATH rehabilitation were performed for 30 minutes per time, respectively. The number of intervention was held for about a month, five times a week(a total of 20 times).
  Interventions: Device: Electrical acupuncture; Device: tDCS; Other: NDT-Bobath Rehabilitation
- Acupuncture + sham tDCS + NDT-Bobath Rehabilitation (Active Comparator): Acupuncture, tDCS, and NDT-BOBATH rehabilitation were performed for 30 minutes per time, respectively. The number of intervention was held for about a month, five times a week(a total of 20 times).
  Interventions: Device: Acupuncture; Device: sham tDCS; Other: NDT-Bobath Rehabilitation

INTERVENTIONS:
Device: Electrical acupuncture — Electrical acupuncture (2Hz, 150 μs) once daily (five times a week), for 20 minutes each session, totaling 20 sessions.
  Arms: Electrical acupuncture+ tDCS + NDT-Bobath Rehabilitation
Device: Acupuncture — Electrical acupuncture (no electricity) once daily (five times a week), for 20 minutes each session, totaling 20 sessions.
  Arms: Acupuncture + sham tDCS + NDT-Bobath Rehabilitation
Device: tDCS — tDCS (1mA) once daily (five times a week), for 20 minutes each session, totaling 20 sessions.
  Arms: Electrical acupuncture+ tDCS + NDT-Bobath Rehabilitation
Device: sham tDCS — tDCS (no electricity) once daily (five times a week), for 20 minutes each session, totaling 20 sessions.
  Arms: Acupuncture + sham tDCS + NDT-Bobath Rehabilitation
Other: NDT-Bobath Rehabilitation — NDT-Bobath Rehabilitation once daily (five times a week), for 30 minutes each session, totaling 20 sessions.

SUMMARY:
The purpose of this study is to confirm the convergence effectiveness of on acupuncture of the chinese medicine and the tDCS of the western medicine on motor function for patients with acute stroke compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Those who within 2 weeks or more and 6 months after a stroke diagnosis.
* Those who have a lesion with a cortex or subcortex
* Adults over 19 years old
* Inpatients and outpatients who can mediate for 4 weeks
* Those who can understand and follow the purpose of this study

Exclusion Criteria:

* Those who fall under the exclusion criteria for electrical acupuncture or acupuncture or tDCS
* Those who have a experience about adverse reaction to the existing electrical acupuncture or acupuncture or tDCS
* Those who have major psychiatric diseases such as major depression disorders, schizophrenia, bipolar disorders, and dementia
* A person who judges that it is not appropriate for a researcher to participate in this study

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Korean version of the Fugl-Meyer Assessment Scale(K-FMA) score | Baseline and Week 4
  The FMA is a validated, instrument assessing average motor function of upper and lower extremity. Possible scores range from 0(worst motor function) to 212(best motor function). Change= (Week 4 Score - Baseline Score).
Change of brain activity | Baseline and Week 4
  The fNIRS(functional Near-Infrared Spectroscopy) is a imaged, instrument assessing average brain activity. Change= (Week 4 Score - Baseline Score).

SECONDARY OUTCOMES:
Change of Korean version of Modified Barthel Index(K-MBI) score | Baseline and Week 4
  The MBI is a validated, instrument assessing average level of ADL(activity of daily living). Possible scores range from 0(maximal independence) to 100(minimal independence). Change= (Week 4 Score - Baseline Score).

CONTACTS AND LOCATIONS:
Overall Officials: Young-Il Shin, Dr., Study Director — Pusan National University Yangsan Hospital
Locations (1):
- Pusan national university Yangsan Hospital, Gyeongsang, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No